CLINICAL TRIAL: NCT06385002
Title: Effect of Combined Administration of Sevoflurane and Remimazolam on Emergence in Patients Undergoing Gynecological Laparoscopic Surgery Under General Anesthesia: a Prospective Randomized Controlled Study
Brief Title: Effect of Combined Administration of Sevoflurane and Remimazolam on Emergence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Assistant professor for fund, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2024-0158
Record Dates: First submitted 2024-04-19; First posted 2024-04-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Gynecological Surgery
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sevoflurane group, S group (No Intervention): The control group will maintain oxygen-air (O2-Air) at 2 L/min and adjust the concentration of sevoflurane to maintain the depth of anesthesia with a bispectral index (BIS) of 40-60.
- Remimazolam/Sevoflurane group, RS group (Active Comparator): After tracheal intubation, the experimental group will maintain oxygen-air (O2-Air) at 2 liters/minute, and remimazolam will be infused at 1.0mg/kg/h, while adjusting the concentration of sevoflurane to maintain the depth of anesthesia with a bispectral index (BIS) of 40-60.
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — After tracheal intubation, the experimental group will maintain oxygen-air (O2-Air) at 2 liters/minute, and remimazolam will be infused at 1.0mg/kg/h, while adjusting the concentration of sevoflurane to maintain the depth of anesthesia with a bispectral index (BIS) of 40-60.
  Other Names: Byfavo
  Arms: Remimazolam/Sevoflurane group, RS group

SUMMARY:
Enhanced recovery after surgery (ERAS) protocols are being explored to improve patient outcomes. The method of inducing anesthesia and maintenance using inhalation anesthetics is common but may delay recovery. Remimazolam, a benzodiazepine-class drug, is noted for its rapid metabolism and fewer hemodynamic changes. Research suggests combining sevoflurane and propofol for anesthesia in adults enhances recovery, while studies in pediatric patients indicate a reduction in emergence agitation with remimazolam. However, the impact of combining sevoflurane and remimazolam on postoperative recovery in adult patients undergoing gynecologic and laparoscopic surgery is not yet studied. The study aims to compare the time to emergence from anesthesia and tracheal extubation between concurrent sevoflurane and remimazolam administration versus sevoflurane alone.

DETAILED DESCRIPTION:
* Laparoscopic oophorectomy or hysterectomy is a commonly performed gynecological surgery, and rapid recovery, pain management, prevention of postoperative nausea and vomiting are important factors determining early discharge and patient satisfaction. With the recent emergence of enhanced recovery after surgery (ERAS), various clinical studies are being conducted to improve the quality of patient recovery through decisions regarding anesthesia methods and agents, fluid administration, prevention of nausea and vomiting, and pain management during surgery.
* The method of inducing anesthesia with intravenous injection of anesthetic agents such as propofol followed by maintenance of anesthesia using inhalation anesthetics is generally performed as a method of general anesthesia. Inhalation anesthetics commonly used for maintenance of anesthesia can be easily administered and removed via ventilation, and they have the advantage of maintaining anesthesia depth relatively easily by monitoring parameters such as bispectral Index (BIS) and end-tidal gas concentration. However, it has the disadvantage of delaying recovery and increasing hospital stay due to postoperative nausea and vomiting, and it decreases average arterial pressure proportionally to the dose due to systemic vasodilation.
* Remimazolam (Byfavo Inj., Hana Pharm Col, Ltd., Seoul, Korea) is a benzodiazepine-class drug used for induction and maintenance of general anesthesia and for sedation during procedures. When remimazolam is used as a general anesthetic, it is rapidly metabolized by enzymes in the liver compared to propofol, resulting in a short context-sensitive half-life of 7.5 minutes and allowing for reversal with flumazenil. Additionally, it is known to induce fewer hemodynamic changes.
* There is research indicating that combining sevoflurane and propofol (target plasma concentration 1.2 mcg/mL) for general anesthesia in adult patients reduces arousal excitement and provides rapid recovery. However, in general anesthesia using desflurane or remimazolam, the time to tracheal extubation was longer in the remimazolam group. Furthermore, there is research suggesting that combining remimazolam with inhalation anesthesia during general anesthesia in pediatric patients can reduce the occurrence of emergence agitation after surgery, but the time to emergence is longer. However, there is currently no research on the effects of combining sevoflurane and remimazolam for general anesthesia in adult patients on postoperative arousal and recovery.

The objective of this study is to investigate whether there is a difference in the time to emergence from anesthesia and time to tracheal extubation in patients undergoing gynecologic and laparoscopic surgery under general anesthesia, comparing the concurrent administration of sevoflurane and remimazolam with the maintenance of anesthesia using sevoflurane alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 19 to 70 undergoing gynecologic and laparoscopic surgery under general anesthesia
* Patients classified as American Society of Anesthesiologists (ASA) physical status classification I or II

  * According to the American Society of Anesthesiologists (ASA) physical status classification:

Class I - Healthy patients without systemic disease Class II - Patients with mild systemic disease without functional limitation Class III - Patients with severe systemic disease that limits activity but is not incapacitating Class IV - Patients with incapacitating systemic disease that is a constant threat to life Class V - Moribund patients who are not expected to survive without the operation Class VI - Brain-dead patients for organ donation

Exclusion Criteria:

* Patients classified as ASA physical status classification III or above
* Pregnant women
* Patients with hypersensitivity to sevoflurane or other halogenated anesthetics, malignant hyperthermia, or a history of it in the patient or family
* Patients with preoperative impairment of consciousness or coma
* Patients undergoing emergency surgery or those who are hemodynamically unstable preoperatively
* Patients with a history of neuromuscular disorders or medication affecting neuromuscular function
* Patients who have taken sedatives (anxiolytics, hypnotics, antipsychotics, antidepressants, or sleeping pills) within 24 hours
* Patients receiving long-term benzodiazepine therapy
* Patients with alcohol or substance dependence
* Patients with allergy history to benzodiazepines or flumazenil
* Patients with genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* Patients with severe hypersensitivity reactions to dextran 40
* Patients with chronic renal failure requiring hemodialysis
* Patients with a history of acute angle-closure glaucoma

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
time to emergence | Immediate after the end of general anesthesia
  A comparison will be made between the time to emergence from anesthesia in patients receiving concurrent administration of sevoflurane and remimazolam versus those maintained on sevoflurane alone after surgery.
time to tracheal extubation | Immediate after the end of general anesthesia
  A comparison will be made between the time to tracheal extubation in patients receiving concurrent administration of sevoflurane and remimazolam versus those maintained on sevoflurane alone after surgery.

SECONDARY OUTCOMES:
usage of vasopressors | During general anesthesia
  usage of vasopressors during general anesthesia
severity of cough | immediate after the end of general anesthesia
  severity of cough during tracheal extubation
time to discharge from the recovery room | immediate after entering the PACU until until achieving post-anesthesia recovery score of 9 or more
  time to discharge from the recovery room
postoperative pain scores | Immediate after entering the PACU, 15 minutes after entering the PACU
  Visual analog scale (VAS) is going to be measured after entering the PACU. The VAS is a validated, subjective measure for acute and chronic pain. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
scores for postoperative nausea and vomiting | Immediate after entering the PACU, 15 minutes after entering the PACU
  Postoperative nausea was evaluated by means of a classical VAS (0-10 cm) device and a 4-point VDS (verbal descriptive scale,0=no nausea, 1=mild, 2=moderate, 3=severe).

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, MD, PhD, Principal Investigator — Department of Anesthesia and Pain Medicine, School of Medicine, Pusan National University
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea